CLINICAL TRIAL: NCT07034482
Title: Efficacy and Safety of Combination Therapy of Intralesional 5-Fluorouracil and Triamcinolone Acetonide in Treatment of Keloids and Hypertrophic Scars: A Prospective Study
Brief Title: Efficacy and Safety of Intralesional 5-Fluorouracil and Triamcinolone Acetonide in Keloids and Hypertrophic Scars
Status: Completed | Type: Observational
Sponsor: Maharajgunj Medical Campus (Other)
Responsible Party: Principal Investigator, Prajjwol Luitel, Principal Investigator, Maharajgunj Medical Campus
Other Study IDs: 54(6-11)E2.077/078
Record Dates: First submitted 2025-06-11; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Keloids
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged 16 years or more, with keloids and HTS's more than 10 mm in size
  Interventions: Drug: Intralesional Triamcinolone 5 mg/ml; Drug: Intralesional 5-fluorouracil

INTERVENTIONS:
Drug: Intralesional Triamcinolone 5 mg/ml — Solution containing 5 mg TAC was injected intralesionally, every week for 6 weeks or until the scar flattened, whichever occurred earlier. Not more than 2 ml of the solution was injected per session, using 27G needle pre-mounted on an insulin syringe.
Drug: Intralesional 5-fluorouracil — Solution containing 45 mg 5-FU was injected intralesionally, every week for 6 weeks or until the scar flattened, whichever occurred earlier. Not more than 2 ml of the solution was injected per session, using 27G needle pre-mounted on an insulin syringe.

SUMMARY:
Pathological scars like keloids and hypertrophic scars (HTS's) cause significant aesthetic, symptomatic and psychological issues to patients. Treatment is challenging with no universally accepted "gold standard" method. Plethora of options is in practice: intralesional (IL) injections, silicon sheets, lasers, cryotherapy, radiotherapy and surgery. This study analysed the effect of combination therapy of IL 5-fluorouracil (5-FU) and triamcinolone acetonide (TAC) in keloids and HTS's.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 years or more, with keloids or hypertrophic scar more than 10 mm in size

Exclusion Criteria:

* Signs of systemic or local infection
* who underwent treatment for same scar in the past 6 months
* Renal failure or liver dysfunction or bone marrow suppression

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study was conducted in the Department of Plastic Surgery and Burns, Tribhuvan University Teaching Hospital, Kathmandu, Nepal, from September 2020 to September 2021. Eligible participants included patients presenting with keloids or hypertrophic scars who met the predefined inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Scar Height | 12 months
  Change in scar height measured in millimeters (mm) using a standardized caliper.
Vancouver Scar Scale (VSS) Score | 12 months
  Change in scar severity based on the Vancouver Scar Scale, a validated tool assessing vascularity, pigmentation, pliability, and height. Scale Range: 0 (normal skin) to 13 (worst scarring)
Patient-Reported Pain Score | 12 months
  Self-reported scar-associated pain using a 10-point Visual Analog Scale (VAS). Scale Range: 0 (no pain) to 10 (worst imaginable pain)
Patient-Reported Pruritus Score | 12 months
  Self-reported itch severity related to the scar, measured using a 10-point Visual Analog Scale (VAS).
  Scale Range: 0 (no itch) to 10 (worst imaginable itch)
Patient-Reported Scar Appearance Score | 12 months
  Self-reported perception of scar appearance using a 10-point Visual Analog Scale (VAS).
  Scale Range: 0 (no visible scar) to 10 (worst possible scar appearance)

CONTACTS AND LOCATIONS:
Overall Officials: Prajjwol Luitel, Principal Investigator — Institute Of Medicine (IOM), Maharajgunj Medical Campus
Locations (1):
- Maharajgunj Medical Campus, Institute of Medicine, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No